CLINICAL TRIAL: NCT05552157
Title: A Phase II/III Multicenter Randomized, Double-Blind, Placebo-Controlled, Two-Stage Adaptive Design, Platform Trial of Investigational Treatments for Primary Prevention of Disease Progression in Dominantly Inherited Alzheimer's Disease
Brief Title: A Study of Potential Disease Modifying Treatments in Individuals at Risk for or With a Type of Early Onset AD Caused by a Genetic Mutation
Acronym: DIAN-TU
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Alzheimer's Association (Other); Eli Lilly and Company (Industry); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DIAN-TU-002 (Master); 5U01AG059798 (NIH)
Record Dates: First submitted 2022-09-19; First posted 2022-09-23 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Alzheimers Disease; Dementia; Alzheimers Disease, Familial
Keywords: Alzheimer's; Alzheimer's Disease; Dementia; Mutation; Genetic Mutation; Dominantly Inherited Alzheimer's Disease; Dominantly Inherited Alzheimer Network; Autosomal Dominant Alzheimer's Disease; Early Onset Alzheimer's Disease; DIAN; DIAN-TU; DIAN TU; DIAD
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Intervention Model Description: Stage 1: Interventional/matching placebo; Stage 2: Open Label Potential for future interventions to be added
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Stage 1: Remternetug (Experimental): Active Remternetug- blinded
  Interventions: Drug: Remternetug (SC)
- Stage 1: Matching Placebo (Remternetug) (Placebo Comparator): Matching placebo
  Interventions: Drug: Matching Placebo (Remternetug)
- Stage 2: Remternetug Open Label (Active Comparator): Open label will start after last dose of Stage 1
  Interventions: Drug: Remternetug (SC)

INTERVENTIONS:
Drug: Remternetug (SC) — Administered subcutaneously every 12 weeks
  Arms: Stage 1: Remternetug; Stage 2: Remternetug Open Label
Drug: Matching Placebo (Remternetug) — Administered as subcutaneous injection of placebo every 12 weeks
  Arms: Stage 1: Matching Placebo (Remternetug)

SUMMARY:
The purpose is to evaluate the biomarker effect, safety, and tolerability of investigational study drugs in participants who are known to have an Alzheimer's disease (AD)-causing mutation. Stage 1 will determine if treatment with the study drug prevents or slows the rate of amyloid beta (Aβ) pathological disease accumulation demonstrated by Aβ positron emission tomography (PET) imaging. Stage 2 will evaluate the effect of early Aβ plaque reduction/prevention on disease progression by assessing downstream non-Aβ biomarkers of AD (e.g., CSF total tau, p-tau, NfL) compared to an external control group from the DIAN-OBS natural history study and the DIAN-TU-001 placebo-treated participants.

DETAILED DESCRIPTION:
This study will recruit participants from the Dominantly Inherited Alzheimer Network observational study (DIAN-OBS), a multicenter international study supported by the National Institutes of Health (Grant Number U01-AG032438; RJ Bateman), Dominantly Inherited Alzheimer Network Trials Unit (DIAN-TU) sites, DIAN-TU partner sites, DIAN Expanded Registry (DIAN-EXR), and families identified by the sites. As part of the DIAN-TU-002 protocol, participants undergo longitudinal assessments that include clinical assessment, cognitive testing, magnetic resonance imaging (MRI) and amyloid imaging, and analysis of cerebrospinal fluid (CSF).

Participants in DIAN are recruited from families that have at least one member who has been identified as having a mutation linked to dominantly inherited Alzheimer's disease (DIAD). The mutations in presenilin 1 (PSEN1), presenilin 2 (PSEN2) and amyloid precursor protein (APP) genes that are associated with DIAD have very high penetrance (near 100%). This study will enroll individuals who are either known to have a known disease-causing mutation, or who are at risk for such a mutation (the child or sibling of a proband with a known mutation) and unaware of their genetic status. Because the age at onset of cognitive changes is relatively consistent within each family and for each mutation, an age at onset is determined for each affected parent or mutation as part of the DIAN-OBS study protocol. This study will enroll participants who are asymptomatic and are within a specific window of time of expected age at onset for their family and/or mutation.

The ability to identify individuals destined to develop Alzheimer's disease (AD) with a high degree of confidence provides a unique opportunity to assess the efficacy of therapies at asymptomatic and very early stages of dementia. Families with known disease-causing mutations are extremely rare and are geographically dispersed throughout the world. These constraints necessitate a specialized study design. Participants in this study will not yet have developed any symptoms of AD; they will be "asymptomatic" carriers of mutations that cause DIAD and would be expected to perform normally on standard cognitive and functional testing. Further, most mutation carriers will have levels of AD-associated amyloid beta (Aβ) and non-Aβ biomarkers that are the same as non-carriers. Imaging and fluid biomarkers will be used to demonstrate that the treatment compounds have engaged their therapeutic targets. A set of cognitive measures designed to assess the very earliest and most subtle cognitive changes will be collected. However, the goal of this study is to address whether decreasing plaque prone Aβ peptides in the absence of measurable or mild elevations of Aβ plaques in participants with minimal to no amyloid plaque at baseline can lead to the subsequent prevention of non-Aβ biomarkers of disease progression. Additionally, because many at-risk individuals decide not to know whether they have the disease-associated mutation, some of the at-risk individuals enrolled in this study will not have the disease-causing mutations; they will be "mutation-negative." It is important to enroll these participants to avoid coercion (e.g., potential participants may feel pressured into genetic testing to learn their genetic status to be eligible for the trial). These mutation-negative individuals will be assigned to the placebo group and data will be used to determine normal ranges of outcome. Participants and site study staff will remain blinded as to these individuals' active or placebo group assignment and mutation status. Thus, the study will be blinded for placebo and for mutation status, except for mutation carriers who are aware of their genetic status. There may be exceptional circumstances as required by local regulation or health authorities where enrollment may be restricted to mutation carriers only, but such mandates will be thoroughly documented and agreed upon by the governing regulatory agency and the study sponsor.

This study is an adaptive-platform-based study. Several different therapies (each referred to as a study drug arm) may be tested in order to increase the likelihood that an effective treatment will be discovered. The compounds are selected for this trial based on mechanism of action and available data on efficacy and safety profile. In the case of multiple study arms, the study design includes a pooled placebo group (referred to as the mutation positive placebos) shared by all study drug arms. Mutation carriers will be assigned to a study drug arm and subsequently randomized within that arm in an overall 1:1 ratio to active drug: placebo. Mutation-negative participants will all receive placebo treatment. Participants and study staff will not be blinded as to which study drug arm each participant has been assigned; they will be blinded to whether participants have been randomized to receive active drug or placebo.

The study has 2 treatment periods: Stage 1 is a blinded placebo-controlled period that will continue until the last randomized participant completes 4 years of treatment (i.e., a common close design), and Stage 2 is an open-label period of 4 years (with a planned 2-year interim efficacy analysis) in which all mutation carriers will receive active drug. At the start of Stage 2, participants who were randomized to placebo in Stage 1 will follow the same dose titration schedule and MRI safety schedule used in Stage 1. Participants who were randomized to active drug in Stage 1 will follow a mock dose titration and will have the same MRI safety schedule used during the initial drug titration as Stage 1 but will remain on the dose that they were on at the end of Stage 1. This will protect the blind to the original treatment assignment from Stage 1. Participants, investigators, and the sponsor's clinical team will remain blinded throughout the study to the Stage 1 treatment assignment.

Stage 1 of the study is designed to test whether the study drug can slow, prevent, or reverse progression of Aβ pathology associated with AD and Stage 2 is designed to assess the study drug's effect on non-amyloid biomarkers of AD that may lead to future slowing or prevention of clinical symptoms of dementia.

Biomarker, cognitive, and/or clinical endpoints will be specified for each study drug arm. Biomarker data will be analyzed for pre-specified endpoints consistent with the drug's mechanism of action and other AD biomarker outcomes. The clinical and cognitive assessments are designed to assess subtle cognitive changes that may be detectable before the onset of dementia as well as cognitive and clinical decline in symptomatic groups.

Roche announced a decision to discontinue most of the company's global trials of gantenerumab. The DIAN-TU has paused the DIAN-TU-002 Primary Prevention Trial related to gantenerumab while considering other potential options for this platform trial.

The DIAN-TU has re-launched the DIAN-TU-002 Primary Prevention Trial with remternetug in collaboration with Eli Lilly and Company as part of this Master Protocol. The remternetug arm is posted under NCT06647498.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent, signed, and dated by the participant and study partner, or by the participant's legally authorized representative if applicable, according to local regulations for the ICF and, if applicable, country specific ICFs.
2. Participant is at least 18 years old.
3. People of childbearing potential

   1. Must have a negative serum pregnancy test at screening (V1)
   2. Must agree not to try to become pregnant during the study until 5 half-lives after the last dose of any study drug.
   3. Must agree not to breastfeed from the time of signed ICF until 5 half-lives after the last dose of any study drug.
   4. If partner is not sterilized, must agree to use highly effective contraceptive measuresfrom screening (V1) until 5 half lives after last dose of any study drug
4. Mutation status :

   1. Participant is a carrier of a mutation in an APP, PSEN1, or PSEN2 gene that is associated with DIAD or does not know their mutation status and there is a mutation in their family pedigree that puts them at a direct risk of inheriting the known mutation;
   2. Participant is -25 to -11 years from predicted age of cognitive symptom onset based on their mutation type or family pedigree Note: If the at-risk parent is deemed a non-carrier through confirmed genetic testing at any time during the study, the participant will be withdrawn.
5. Cognitive status of participant is normal (CDR-SB 0).
6. Fluency in DIAN-TU trial approved language and evidence of adequate premorbid intellectual functioning. Participants must be fluent in languages for which cognitive and clinical measures have been translated and validated for use in the DIAN-TU. Fluency is generally defined as daily or frequent functional use of a language generally from birth or a young age. In cultures where multiple languages are spoken or for participants who are multilingual, determination as to whether a participant's level of fluency in languages for which clinical and cognitive measures are available meets qualification for the study should be made by the site PI.
7. Participant has adequate visual and auditory abilities to perform all aspects of the cognitive and clinical assessments.
8. Participant is receiving stable doses of medication(s) for the treatment of non-excluded medical condition(s) for at least 30 days prior to baseline visit (V2) except for medications taken for episodic conditions (e.g., migraine abortive therapy, antibiotics, and other medications for upper respiratory and gastrointestinal ailments).
9. The participant has a study partner who in the PI's judgment can provide accurate information as to the participant's cognitive and functional abilities, who agrees to provide information at the study visits that require study partner input for scale completion, and who signs the necessary ICF, if applicable.
10. The participant agrees not to donate blood or blood products for transfusion from the time of Screening (V1) for a study drug arm, for the duration of the study, and for 5 half lives after the final dose of study drug.
11. In the opinion of the PI, the participant will be compliant and have a high probability of completing the study.
12. The participant is able and willing to complete all study-related testing, evaluations, and procedures.

Exclusion Criteria:

1. Significant neurologic disease (other than AD) or psychiatric disease that may currently or during the study affect cognition or the participant's ability to complete the study. This would include disorders such as: recent or severe head trauma causing cognitive change, seizure disorder, neurodegenerative disease other than DIAD, hydrocephalus, cerebral/spinal hematoma, inflammatory disease, CNS infection (e.g., encephalitis or meningitis), neoplasm, toxic exposure, metabolic disorder (including hypoxic or hypoglycemic episodes) or endocrine disorder; psychiatric disorders such as schizophrenia, schizoaffective disorder, bipolar disorder or major depression, or any other psychiatric condition/disorder which could significantly interfere with the participant's cooperative participation (e.g., prominent anxiety, agitation or behavioral problems). Disorders that are controlled medically or remote history of these disorders (e.g., history of febrile seizures in childhood) that are not likely to interfere with cognitive function and compliance with study procedures are not exclusionary.
2. At high risk for suicide, e.g., significant suicidal ideation or attempt within last 12 months, current major depression (as defined in Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition [DSM-V]), or increased suicide risk based on screening Columbia Suicide Severity Rating Scale (C-SSRS). Current stable mild depression or current use of antidepressant medications are not exclusionary.
3. History of clinically evident stroke or history of clinically important carotid or vertebrobasilar stenosis, plaque, or other prominent risk factor for stroke or cerebral hemorrhage (including atrial fibrillation and anticoagulation, documented transient ischemic attack [TIA] in the last 12 months) that may be interfering with cognition or is likely to impact with the participant's ability to complete the study. Low dose aspirin (≤ 325 mg daily) is not exclusionary.
4. Alcohol or substance use sufficient to meet DSM-V criteria currently or within the past year.
5. History of or Baseline (V2) visit brain MRI scan indicative of any other significant abnormality, definite microhemorrhages, evidence of a cerebral contusion, encephalomalacia, or aneurysms. Minor or clinically insignificant imaging findings are not exclusionary.
6. Presence of certain implanted medical devices, such as some pacemakers, aneurysm clips, artificial heart valves, ear implants, or foreign metal objects in the eyes, skin, or body which would preclude MRI scan.
7. Cardiovascular complications such as uncontrolled hypertension, history of myocardial infarcts, heart failure, atrial fibrillation, long QT interval on ECG likely to interfere with participation in or analysis of the trial in the opinion of the investigator
8. Hepatic or renal abnormalities that in the opinion of the investigator would interfere with participation in or analysis of the trial.
9. History of Human Immunodeficiency Virus (HIV) infection, history of Hepatitis B infection within the past year, history of Hepatitis C infection which has not been adequately treated or history of spirochete infection (e.g., syphilis, Lyme) of the CNS, or history of other infection with high risk for interfering with participation or interpretation of the study in the opinion of the investigator.
10. History of clinically significant multiple or severe drug allergies, significant atopy, or severe post-treatment hypersensitivity reactions (including but not limited to erythema multiforme major, linear IgA dermatosis, toxic epidermal necrolysis, and/or exfoliative dermatitis) or sensitivity to study-drug specific PET imaging agents with a high risk for interfering with participation or interpretation of the study in the opinion of the investigator.
11. Treatment with immunosuppressive medications (e.g., systemic corticosteroids) within 90 days prior to Baseline (V2) visit (topical and nasal corticosteroids and inhaled corticosteroids for asthma are permitted) or chemotherapeutic agents for malignancy within the last 3 years.
12. Current clinically significant abnormalities of thyroid function, or clinically significant deficiency in vitamin B12. Vitamin B12 less than the lower limits of normal with normal methylmalonic acid (MMA)/homocysteine is not deemed clinically significant, therefore not exclusionary.
13. Unstable or poorly controlled diabetes which the investigator believes may interfere with participation in or analysis of the study protocol. Participants may be rescreened after 3 months to allow optimization of diabetic control
14. Morbid obesity with significant comorbidities or that would preclude MRI imaging.
15. Current use of anticoagulants (e.g., warfarin, dabigatran, rivaroxaban, or apixaban). Daily use of low dose (< 325 mg) aspirin is not exclusionary.
16. Have been exposed to a monoclonal antibody targeting Aβ peptide within the past 6 months or 5 half-lives from screening, whichever is longer.
17. Received any other investigational pharmacological treatment within 3 months of Screening or 5 half-lives, whichever is longer.

    Note: Use of approved treatments for AD and other medications may be permitted in this study.
18. Lack of sufficient venous access.
19. Clinically relevant abnormalities in hematology, coagulation, or clinical chemistry.
20. History of cancer that the investigator believes has high risk of recurrence and impacting study participation or analysis.
21. Any other medical condition that could be expected to progress, recur, or change to such an extent that it could bias the assessment of the clinical or mental status of the participant to a significant degree or put the participant at special risk.
22. Currently, or within the last month prior to screening, participated in a clinical study, including a nonpharmacological study, without prior approval.
23. Participants with the "Dutch" APP E693Q mutation.
24. Unable to complete baseline visit (V2) procedures with appropriate cognitive and clinical scores for eligibility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2034-03-30 (Estimated); Study Completion 2034-08-30 (Estimated)

PRIMARY OUTCOMES:
Stage 1: Evaluate the ability of study drug to prevent or slow the rate of Aβ accumulation compared with placebo in participants with mutations that cause DIAD | Baseline and Week 208
  Defined in each drug-specific appendix; will be an assessment of biomarkers of early-stage disease (e.g., amyloid PET, soluble amyloid, soluble phospho-tau) compared with baseline in each treatment group
Stage 2: Evaluate the effect of anti-amyloid treatment on downstream biomarkers of AD | Stage 2 Week 208
  If applicable, will be defined in each drug-specific appendix, and will be an assessment of the change in progression of biomarkers representing tau, neurodegenerative, and inflammatory pathobiological events in the disease cascade for temporally different periods of the pre-symptomatic phases of the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Eric M McDade, DO, Study Director — Washington University School of Medicine
Locations (35):
- United States (12):
  - University of Alabama in Birmingham, Birmingham, Alabama
  - University of California San Diego Medical Center, La Jolla, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Washington University in St. Louis, St Louis, Missouri
  - New York University Medical Center, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Butler Hospital, Providence, Rhode Island
  - Kerwin Research and Memory Center, Dallas, Texas
  - University of Washington, Seattle, Washington
- Instituto de Investigaciones Neurologicas Raul Carrea, FLENI, Ciudad Autonoma de Buenos Aire, Argentina
- Australia (2):
  - Neuroscience Research Australia, Randwick, New South Wales
  - Mental Health Research Institute, Melbourne, Victoria
- Canada (4):
  - UBC Hospital, Vancouver, British Columbia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - McGill Center for Studies in Aging, Verdun, Quebec
  - CHU de Quebec - Hôpital de l' Enfant Jésus, Québec
- Grupo de Neurociencias Sede de la Universidad de Antioquia, Medellín, Colombia
- France (5):
  - CHU de Toulouse - Hôpital Purpan, Toulouse, Haute Garonne
  - Hopital Roger Salengro - CHU Lille, Lille, Nord
  - Groupe Hospitalier Pitie-Salpetriere, Paris, Paris
  - Hopital Neurologique Pierre Wertheimer, Bron, Rhone
  - CHU de Rouen - Hôpital Charles Nicolle, Rouen, Seine Maritime
- Germany (2):
  - Universitaetsklinikum Tubingen, Tübingen, Baden-Wurttemberg
  - LMU-Campus Grosshadern, Munich, Bavaria
- Italy (2):
  - IRCCS Centro San Giovanni di Dio Fatebenefratelli, Brescia
  - Azienda Ospedaliera Universitaria Careggi, Florence
- Instituto Nacional de Neurologia y Neurocirugia Manuel Velasco Suarez, Mexico City, Mexico City, Mexico
- Brain Research Center, Amsterdam, Netherlands
- New Zealand Brain Research Institute, Christchurch, New Zealand
- University of Puerto Rico, School of Medicine, San Juan, Puerto Rico, Puerto Rico
- Hospital Clínic I Provincial de Barcelona, Barcelona, Barcelona, Spain
- The National Hospital for Neurology and Neurosurgery, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Access to DIAN-TU trial data will follow the DIAN-TU data access policy, which complies with the guidelines established by the Collaboration for Alzheimer's Prevention [CAP REF].

REFERENCES:
- [Background] McDade E, Wang G, Gordon BA, Hassenstab J, Benzinger TLS, Buckles V, Fagan AM, Holtzman DM, Cairns NJ, Goate AM, Marcus DS, Morris JC, Paumier K, Xiong C, Allegri R, Berman SB, Klunk W, Noble J, Ringman J, Ghetti B, Farlow M, Sperling RA, Chhatwal J, Salloway S, Graff-Radford NR, Schofield PR, Masters C, Rossor MN, Fox NC, Levin J, Jucker M, Bateman RJ; Dominantly Inherited Alzheimer Network. Longitudinal cognitive and biomarker changes in dominantly inherited Alzheimer disease. Neurology. 2018 Oct 2;91(14):e1295-e1306. doi: 10.1212/WNL.0000000000006277. Epub 2018 Sep 14. PMID 30217935
- [Background] Mills SM, Mallmann J, Santacruz AM, Fuqua A, Carril M, Aisen PS, Althage MC, Belyew S, Benzinger TL, Brooks WS, Buckles VD, Cairns NJ, Clifford D, Danek A, Fagan AM, Farlow M, Fox N, Ghetti B, Goate AM, Heinrichs D, Hornbeck R, Jack C, Jucker M, Klunk WE, Marcus DS, Martins RN, Masters CM, Mayeux R, McDade E, Morris JC, Oliver A, Ringman JM, Rossor MN, Salloway S, Schofield PR, Snider J, Snyder P, Sperling RA, Stewart C, Thomas RG, Xiong C, Bateman RJ. Preclinical trials in autosomal dominant AD: implementation of the DIAN-TU trial. Rev Neurol (Paris). 2013 Oct;169(10):737-43. doi: 10.1016/j.neurol.2013.07.017. Epub 2013 Sep 6. PMID 24016464
- [Background] Bateman RJ, Xiong C, Benzinger TL, Fagan AM, Goate A, Fox NC, Marcus DS, Cairns NJ, Xie X, Blazey TM, Holtzman DM, Santacruz A, Buckles V, Oliver A, Moulder K, Aisen PS, Ghetti B, Klunk WE, McDade E, Martins RN, Masters CL, Mayeux R, Ringman JM, Rossor MN, Schofield PR, Sperling RA, Salloway S, Morris JC; Dominantly Inherited Alzheimer Network. Clinical and biomarker changes in dominantly inherited Alzheimer's disease. N Engl J Med. 2012 Aug 30;367(9):795-804. doi: 10.1056/NEJMoa1202753. Epub 2012 Jul 11. PMID 22784036
- [Background] Navitsky M, Joshi AD, Kennedy I, Klunk WE, Rowe CC, Wong DF, Pontecorvo MJ, Mintun MA, Devous MD Sr. Standardization of amyloid quantitation with florbetapir standardized uptake value ratios to the Centiloid scale. Alzheimers Dement. 2018 Dec;14(12):1565-1571. doi: 10.1016/j.jalz.2018.06.1353. Epub 2018 Jul 11. PMID 30006100
- [Background] Demattos RB, Lu J, Tang Y, Racke MM, Delong CA, Tzaferis JA, Hole JT, Forster BM, McDonnell PC, Liu F, Kinley RD, Jordan WH, Hutton ML. A plaque-specific antibody clears existing beta-amyloid plaques in Alzheimer's disease mice. Neuron. 2012 Dec 6;76(5):908-20. doi: 10.1016/j.neuron.2012.10.029. PMID 23217740
- [Background] Young AL, Oxtoby NP, Daga P, Cash DM, Fox NC, Ourselin S, Schott JM, Alexander DC; Alzheimer's Disease Neuroimaging Initiative. A data-driven model of biomarker changes in sporadic Alzheimer's disease. Brain. 2014 Sep;137(Pt 9):2564-77. doi: 10.1093/brain/awu176. Epub 2014 Jul 9. PMID 25012224
- [Background] McDade E, Bateman RJ. Tau Positron Emission Tomography in Autosomal Dominant Alzheimer Disease: Small Windows, Big Picture. JAMA Neurol. 2018 May 1;75(5):536-538. doi: 10.1001/jamaneurol.2017.4026. No abstract available. PMID 29435570
- [Background] Wang G, Berry S, Xiong C, Hassenstab J, Quintana M, McDade EM, Delmar P, Vestrucci M, Sethuraman G, Bateman RJ; Dominantly Inherited Alzheimer Network Trials Unit. A novel cognitive disease progression model for clinical trials in autosomal-dominant Alzheimer's disease. Stat Med. 2018 Sep 20;37(21):3047-3055. doi: 10.1002/sim.7811. Epub 2018 May 14. PMID 29761523
- [Background] Weninger S, Carrillo MC, Dunn B, Aisen PS, Bateman RJ, Kotz JD, Langbaum JB, Mills SL, Reiman EM, Sperling R, Santacruz AM, Tariot PN, Welsh-Bohmer KA. Collaboration for Alzheimer's Prevention: Principles to guide data and sample sharing in preclinical Alzheimer's disease trials. Alzheimers Dement. 2016 May;12(5):631-2. doi: 10.1016/j.jalz.2016.04.001. No abstract available. PMID 27157073
- [Background] Grill JD, Bateman RJ, Buckles V, Oliver A, Morris JC, Masters CL, Klunk WE, Ringman JM; Dominantly Inherited Alzheimer's Network. A survey of attitudes toward clinical trials and genetic disclosure in autosomal dominant Alzheimer's disease. Alzheimers Res Ther. 2015 Jul 22;7(1):50. doi: 10.1186/s13195-015-0135-0. eCollection 2015. PMID 26203303
- [Background] McDade E, Bateman RJ. Stop Alzheimer's before it starts. Nature. 2017 Jul 12;547(7662):153-155. doi: 10.1038/547153a. No abstract available. PMID 28703214
- [Background] Ryman DC, Acosta-Baena N, Aisen PS, Bird T, Danek A, Fox NC, Goate A, Frommelt P, Ghetti B, Langbaum JB, Lopera F, Martins R, Masters CL, Mayeux RP, McDade E, Moreno S, Reiman EM, Ringman JM, Salloway S, Schofield PR, Sperling R, Tariot PN, Xiong C, Morris JC, Bateman RJ; Dominantly Inherited Alzheimer Network. Symptom onset in autosomal dominant Alzheimer disease: a systematic review and meta-analysis. Neurology. 2014 Jul 15;83(3):253-60. doi: 10.1212/WNL.0000000000000596. Epub 2014 Jun 13. PMID 24928124
- [Background] Weng H, Bateman R, Morris JC, Xiong C. Validity and power of minimization algorithm in longitudinal analysis of clinical trials. Biostat Epidemiol. 2017;1(1):59-77. doi: 10.1080/24709360.2017.1331822. Epub 2017 Jun 13. PMID 29250611
- See also: Expanded registry — http://www.dianexr.org/